CLINICAL TRIAL: NCT05674383
Title: Ultrasound-guided Axillary Nerve Block Trial
Brief Title: Ultrasound Guided Axillary Nerve Block Compared to Hematoma Block in Patients With Closed Reposition of Distal Forearm Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, Bram Rook, Investigator, Frisius Medisch Centrum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL75603.099.20.
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Distal Radius Fracture; Forearm Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive an axillary plexus nerve block as pain reduction before the fracture repositioning.
  Interventions: Procedure: Axillary plexus nerve block
- Control group (Active Comparator): The control group will receive a fracture hematoma block as pain reduction before the fracture repositioning.
  Interventions: Procedure: Fracture hematoma block

INTERVENTIONS:
Procedure: Axillary plexus nerve block — Axillary plexus nerve block: an ultrasound-guided axillary plexus nerve block with a single injection of lidocaine 1%.
  Arms: Intervention group
Procedure: Fracture hematoma block — Fracture hematoma block: a blinded single injection into the fracture with lidocaine 1%.
  Arms: Control group

SUMMARY:
Rationale: For distal forearm fractures the investigators propose an anaesthetic method using an ultrasound guided axillary nerve block (ANB, an established technique) for pain reduction during reposition dislocated fractures. Nowadays a fracture hematoma block (FHB) is common practice, but is suboptimal due to variability between performing physicians and is often experienced as a painful procedure. The investigators want to investigate if ANB is an effective, safe and efficient option in pain reduction in patients of an ED (emergency department) population with a distal forearm fracture.

Objective: To compare ultrasound-guided ANB with FHB for analgesia during reposition of non-operatively treated forearm fractures Study design: A randomized controlled trial. Study population: Patients ≥ 16 years of age with a closed, isolated and displaced distal forearm fracture requiring manipulative reposition.

Intervention (if applicable): The intervention group will receive an ANB on the ipsilateral arm of the fracture. The control group will get a FHB.

Main study parameters/endpoints: The primary outcome is pain score on a 11-point NRS (numeric rating scale) (0-10) during closed reposition of the dislocated distal forearm fracture in both groups. Main endpoint of this study is achieving a reduction of at least 2 points between both groups. This is considered as clinical relevant.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients participating in the research group are believed to have less pain and more comfort during reposition of the dislocated fracture. The investigators expect no other or more complications compared to standard care since the known complications are the same for both infiltrative anaesthetic interventions and are rare. Moreover, both procedures are common practice, therefore potential complications will be taken care of properly. The investigators expect there is no prolonged length of stay in the ED.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the ED with a X-ray confirmed dislocated distal forearm fracture, defined as fracture < 3cm within the radiocarpal joint with an abnormal anatomic position (dorsal angulation >10°, volar angulation >20°, radioulnar inclination <15°, >5mm radial collapse or intra-articular incongruence >2mm.
* ≥ 16 years of age
* Patients who have adequate knowledge and understanding of the Dutch language

Exclusion Criteria:

* 'Open' fractures requiring surgery
* Multi-trauma patients
* Abnormal neurovascular examination requiring immediate reposition or surgery
* Pre-existent osteosynthesis material in situ on the present fracture site.
* Skin injury, local infection or recent burns hindering the use of ultrasound.
* Allergy for local anaesthetics
* Inability to give informed consent (cognitive impairments, no good understanding of the Dutch or English language)
* Severe coagulopathy (i.e. severe thrombocytopenia, haemophilia.). Usage of anticoagulation is not an contra-indication, since any bleeding complication has few adverse consequences(20).
* High risk on compartment syndrome (in consultation with surgery department).

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Pain score | 15 minutes
  The primary outcome is pain measured on a pain score using a 11-point NRS (0-10) during closed reposition of the dislocated distal forearm fracture in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Heleen Lameijer, Dr, Principal Investigator — Heleen.Lameijer1@mcl.nl
Locations (1):
- Medisch centrum Leeuwarden, Leeuwarden, Provincie Friesland, Netherlands

IPD SHARING:
Plan to Share IPD: No